CLINICAL TRIAL: NCT06962085
Title: Effect of Sacral Erector Spinae Plane Block on Postoperative Pain in Transurethral Prostate Resection Surgery
Brief Title: Sacral Erector Spinae Plane Block in Transurethral Prostate Resection Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Adiyaman University (Other)
Responsible Party: Principal Investigator, Fadime Tosun, Assistant Professor, Adiyaman University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ADYU-AR-FT-01
Record Dates: First submitted 2025-04-14; First posted 2025-05-08 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: TURP(Transurethral Resection of Prostate)
Keywords: Bilateral sacral erector spinae plane block; Opioid consumption; Numerical pain scores; Quality of Recovery-15 (QoR-15T); TUR-P
MeSH Terms: interventions — Analgesics, Opioid

STUDY DESIGN:
Intervention Model Description: Two groups as Control and Block groups
Who Masked: Care Provider
Masking Description: Nurses who evaluate the pain score and satisfaction survey during the postoperative follow-up of the patients will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Active Comparator): After general anesthesia is applied, hemodynamic values (noninvasive blood pressure, heart rate, peripheral oxygen saturation) and total remifentanil (Rentanil 2 mg. VEM İlaç San. Ve Tic. A.Ş, İstanbul, Türkiye) use will be recorded during the operation and numerical pain scores and total meperidine (Aldine 100mg/2mL. VEM İlaç San. Ve Tic. A.Ş, İstanbul, Türkiye) use at 0, 2, 4, 6, 12 and 24 hours after the operation will be recorded. At the 24th hour, the Turkish version of the Quality of Recovery-15 (QoR-15T) Questionnaire will be filled out and recorded.
  Interventions: Drug: Opioid Analgesics
- sacral erector spinae plane block group (Active Comparator): In the group where the block will be applied, bilateral sacral erector spinae plane block will be performed with local anesthetic (10 mL 0.25% bupivacaine (Marcaine %0,5. AstraZeneca Ltd, İstanbul, Türkiye)+ 5 mL 1% lidocaine (Lidon 100 mg/ 5mL. ONFARMA İlaç San. Ve Tic. A.Ş, Ankara, Türkiye) after the sacral intermedian crest is visualized with preoperative ultrasound. After general anesthesia is applied, hemodynamic values (noninvasive blood pressure, heart rate, peripheral oxygen saturation) and total remifentanil (Rentanil 2 mg. VEM İlaç San. Ve Tic. A.Ş, İstanbul, Türkiye) use will be recorded during the operation. Additionally, numerical pain scores and total meperidine (Aldine 100mg/2mL. VEM İlaç San. Ve Tic. A.Ş, İstanbul, Türkiye) use at 0, 2, 4, 6, 12 and 24 hours after the operation will be recorded. At the 24th hour, the Turkish version of the Quality of Recovery-15 (QoR-15T) Questionnaire will be filled out and recorded.
  Interventions: Procedure: sacral erector spinae plane block group; Drug: Opioid Analgesics

INTERVENTIONS:
Procedure: sacral erector spinae plane block group — In the block group, bilateral sacral erector spinae plane block (10 mL 0.25% bupivacaine (Marcaine %0,5. AstraZeneca Ltd, İstanbul, Türkiye) + 5 mL 1% lidocaine (Lidon 100 mg/ 5mL. ONFARMA İlaç San. Ve Tic. A.Ş, Ankara, Türkiye) will be performed in the lateral position with the help of ultrasound before surgery.
  Arms: sacral erector spinae plane block group
Drug: Opioid Analgesics — Sacral arrector spine block will not be performed in this group. After general anesthesia, hemodynamic values (noninvasive blood pressure, heart rate, peripheral oxygen saturation) and total remifentanil (Rentanil 2 mg. VEM İlaç San. Ve Tic. A.Ş, İstanbul, Türkiye) use will be recorded during the operation. Additionally, numerical pain scores and total meperidine (Aldine 100mg/2mL. VEM İlaç San. Ve Tic. A.Ş, İstanbul, Türkiye) use at 0, 2, 4, 6, 12 and 24 hours after the operation will be recorded. At the 24th hour, the Turkish version of the Quality of Recovery-15 (QoR-15T) Questionnaire will be filled out and recorded.

SUMMARY:
The aim of this study is to investigate the effects of bilateral sacral erector spinae plane block on hemodynamic values, postoperative pain, analgesic use and patient satisfaction during operative period in Transurethral Prostate Resection surgeries under general anesthesia.

DETAILED DESCRIPTION:
The study included patients who were planned to undergo transurethral prostate resection, were informed about the study, and agreed to participate in the study with their written consent, were over 18 years of age, and were in the ASA I-II risk group. Those who did not agree to participate in the study, patients under 18 years of age, and those in the ASA III-IV risk group were excluded from the study. Patients who agreed to participate in the study were divided into two groups using the sealed envelope method, and general anesthesia was applied to both groups. In the group where the block was to be applied, bilateral sacral erector spinae plane block was performed with local anesthetic (10 mL 0.25% bupivacaine + 5 mL 1% lidocaine) after the 3rd sacral intermedian crest was visualized with preoperative ultrasound. No additional intervention was performed on the patients in the control group other than the surgical procedure and general anesthesia. The hemodynamic values (noninvasive blood pressure, heart rate, peripheral oxygen saturation) of all patients during the operation, total opioid use (remifentanil) during the surgery, and NRS, nausea/vomiting and tramadol amounts at 0, 2, 4, 6, 12, and 24 hours postoperatively were recorded and the values were compared in both groups. Thus, it was aimed to evaluate the effects of sacral erector spinae plane block in transurethral prostate resection operations.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were scheduled for transurethral prostate resection,
* Who agreed to participate in the study,
* Who were over 18 years old
* ASA I-II risk group

Exclusion Criteria:

* Patients who did not agree to participate in the study,
* Those under 18 years old
* ASA III-IV risk group

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Since the patient group undergoing transurethral prostate surgery was male, only male gender was included in the study.
Enrollment: 60 (Actual)
Dates: Start 2024-09-05 (Actual); Primary Completion 2026-01-01 (Actual); Study Completion 2026-01-08 (Actual)

PRIMARY OUTCOMES:
postoperative opioid use | 24 hours
  Opioid use will be recorded at 0, 2, 4, 6, 12 and 24 hours after the operation.

SECONDARY OUTCOMES:
intraoperative opioid use | intraoperative
  Total opioid use (remifentanil) during the operation will be recorded.
numerical pain score | 24 hours
  Postoperatively, numerical pain scores (NRS) will be recorded at 0, 2, 4, 6, 12 and 24 hours and these values will be compared and recorded in both groups. Numerical pain scores (NRS) are the scale used to measure pain intensity. This scale gives a numerical value between 0 and 10, with 0 being 'no pain' and 10 being 'worst imaginable pain'.
QoR-15T (Turkish) quality of recovery scale | 24 hours
  The Quality of Recovery-15 (QoR-15) at 24 hours scale is a patient-reported outcome questionnaire that measures the quality of postoperative recovery. The validity of Quality of Recovery-15 (QoR-15) has been proven in many languages. In our study, the Turkish Quality of Recovery-15 (QoR-15T) will be used to measure postoperative recovery in the Turkish population. The Turkish Quality of Recovery-15 (QoR-15T) scale consists of 2 parts and a total of 15 questions are asked to patients. Patients can score each question between 0 and 10, so the total Turkish Quality of Recovery-15 (QoR-15T) score can range from 0 to 150. A higher score indicates a better recovery quality.

CONTACTS AND LOCATIONS:
Locations (1):
- Adıyaman University Faculty of Medicine Anesthesiology and Reanimation, Merkez, Adıyaman Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No